CLINICAL TRIAL: NCT03701841
Title: Efficacy, Safety and Cost-effectiveness of PEG-rhG-CSF for Primary Prophylaxis Versus Secondary Prophylaxis of Chemotherapy Induced Neutropenia in Patients Receiving Chemotherapy With High-risk FN: a Real World Study
Brief Title: Efficacy, Safety and Cost-effectiveness of PEG-rhG-CSF for Primary vs Secondary Prophylaxis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Yue-Yin Pan, Chief Physician, Anhui Provincial Hospital
Other Study IDs: AHP-PSPRWS
Record Dates: First submitted 2018-09-27; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Chemotherapy-induced Neutropenia
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEG-rhG-CSF primary prophylaxis: Patients receiving chemotherapy who have a overall FN risk >=20% receive PEG-rhG-CSF for primary prophylaxis
  Interventions: Drug: PEG-rhG-CSF
- PEG-rhG-CSF secondary prophylaxis: Patients receiving chemotherapy who had FN or dose-limited neutropenia receive PEG-rhG-CSF for secondary prophylaxis
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF — All patients need to receive PEG-rhG-CSF 6mg approximately 24h or 48h after chemotherapy administration once per cycle, at least 2 cycles

SUMMARY:
This trial is a multicenter, non-interventional, registered real-world clinical study. Based on available evidence and recommendations of guidelines, tumor patients with high risk of FN and eligible for all enrollment criteria were recruited into primary prophylaxis of PEG-rhG-CSF or secondary prophylaxis of PEG-rhG-CSF according to the real-world clinical pathway without randomization. All patients need to receive at least 2 cycles of PEG-rhG-CSF prophylaxis. Researchers will record the incidence of FN, RDI, FN-related hospitalization, antibiotic use, direct medical care and indirect medical care cost under the real clinical conditions, and assess the efficacy, safety and cost-effectiveness of PEG-rhG-CSF primary prophylaxis versus secondary prophylaxis through sub-group analysis and exploratory research.

DETAILED DESCRIPTION:
Patients with cancer planning for chemotherapy assessed with high risk of febrile neutropenia (FN) according to NCCN and ASCO guidelines are recruited, receiving primary or secondary prophylaxis of PEG-rhG-CSF according to real-world clinical pathway in local cancer center for at least 4 cycles of chemotherapy. The primary outcome is the incidence of FN rate and proportion of patients completing chemotherapy on schedule, the second outcomes are the incidence of 3-4 grade of neutropenia, FN-related hospitalization and antibiotic use, incidence of reduction and delay of chemotherapy dose, safety and pharmacoeconomics of PEG-rhG-CSF.

ELIGIBILITY:
Inclusion Criteria:

1. Before the start of the study, all patients have been fully understood the research and the must sign the informed consent
2. Aged 13 years or older
3. accept at least 4 cycles of chemotherapy
4. ECOG PS 0-2
5. expected survival time ≥ 3 months
6. with -high risk of FN according to researchers

Exclusion Criteria:

1. accepted stem cell or bone marrow transplant
2. undergoing any other clinical trial
3. uncontrolled infection, temperature≥38℃
4. per-week scheme chemotherapy
5. severe and uncontrolled diabetes
6. People with allergic diseases or allergies, or who are allergic to this or other genetically engineered Escherichia coli-derived biological products
7. Suspected or confirmed drug use, drug abuse, alcoholics
8. Severe mental or neurological disorders affecting informed consent and/or adverse effect presentation or observation
9. Severe heart, kidney, liver and other important organs chronic diseases
10. Pregnancy or lactation in women or women with gestation detection positive before the first time using drug
11. Patients who have fertility but are unwilling to receive contraception or partners are not willing to accept contraceptives
12. The investigator believes that the patient's condition is not suitable for this clinical study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer planning for chemotherapy assessed with high risk of febrile neutropenia (FN) according to NCCN and ASCO guidelines are recruited, receiving primary or secondary prophylaxis of PEG-rhG-CSF according to real-world clinical pathway in local cancer center for at least 4 cycles of chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of FN rate | through study completion, an average of 2 year
  FN was defined as fever >=38.3°C orally (>=38.0°C for a duration over 2h) or axillary temperature >=38.1°C (>=37.8°C for a duration over 2h) and ANC < 0.5 X 10*9/L
Proportion of patients completing chemotherapy on schedule | through study completion, an average of 2 year
  proportion of patients completing chemotherapy on schedule

SECONDARY OUTCOMES:
Incidence of 3-4 grade of neutropenia | through study completion, an average of 2 year
  the second outcomes are the incidence of 3-4 grade of neutropenia
FN-related hospitalization and antibiotic use | through study completion, an average of 2 year
  FN-related hospitalization and antibiotic use

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincial cancer center, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided